CLINICAL TRIAL: NCT03108950
Title: Dose-Response Effects of Transformative Exercise in Improving Health and Function in Adults With Spinal Cord Injury and Multiple Sclerosis
Brief Title: From Clinic to Community: An Information and Communication Technology (ICT) Home-Based Exercise Training System for Translating Clinical Findings
Acronym: TExT-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Lakeshore Foundation (Other)
Responsible Party: Principal Investigator, James Rimmer, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F160404004
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis; Stroke
MeSH Terms: conditions — Multiple Sclerosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-Based Movement to Music (Experimental): The Movement to Music classes are composed of a set of exercises tailored to the specific needs and capabilities of each target group. The class will consist of and aerobic component and a strength component performed to varying music tempos. All movements will be choreographed by qualified dance instructors. Intervention is delivered using video-conferencing to connect the participant to their instructor.
  Interventions: Behavioral: Movement to Music

INTERVENTIONS:
Behavioral: Movement to Music — The Movement to Music classes are composed of a set of exercises tailored to the specific needs and capabilities of each target group. The class will consist of and aerobic component and a strength component performed to varying music tempos. All movements will be choreographed by qualified dance instructors. Intervention is delivered using video-conferencing to connect the participant to their instructor.
  Other Names: M2M

SUMMARY:
The specific aim of the study in our example is to conduct a feasibility translational home-based exercise trial established in the LEADERS (R2) project with the TExt-ME tele-exercise training system for participants with neurologic disability. We hypothesize that participants in this home-based tele-exercise training program will achieve similar gains in health and function outcomes as the onsite exercise training program. Further, there will be no difference in adverse side effects (safety) between the home-based and onsite exercise treatment groups.

DETAILED DESCRIPTION:
TExT-ME is a home-based tele-exercise study providing a novel exercise program to participants with neurologic disabilities. The exercise curriculum is a Movement 2 Music (M2M) program developed during phase 2 of the grant (clinicaltrials.gov identifier NCT02533882). The exercise exercise classes are taught by trained dance instructors and are composed of a set of exercises tailored to the specific needs and capabilities of adults with neurologic disability. Each set of exercises is performed to high and low tempo music based on the individual's baseline level of function, with adjustments made to increase or decrease intensity if needed. The class consists of several training components: a) warmup (10 min.) to increase range of motion; strength/balance (15-20 min), aerobics (25-30 min. with rest periods as necessary); cool down (5 min).

The TExT-ME training and monitoring system is a user-centered design (UCD) involving a tele-exercise coach (e.g., a trained research staff person) interacting remotely with a participant in their home using video conferencing programs. Participants wear monitors to maintain safe levels of exercise and provide feedback regarding exercise intensity to the instructors. Self-reported indicators of exercise intensity are also collected using rating of perceived exertion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stroke
* MS - mild to moderate disability (Patient Determined Disease Steps Score 0-6)
* Able to use arms or arm/legs for exercise
* Ambulatory or use manual wheelchair

Exclusion Criteria:

* Cognitive impairment (Mini-Mental State Exam score < 24)
* Recent weight change (+/- 25 pounds in 1 year)
* Poorly controlled blood pressure
* Cardiovascular disease event within the past six months
* Severe pulmonary disease
* Renal failure
* Current tobacco user or quit within the last six months
* Current use of medications for psychosis
* Active pressure ulcers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness as measured by sub-maximal VO2 | 12 weeks
  Submax VO2 is assessed by the six minute walk test or the six minute push test. Participants wear a portable metabolic cart while walking or pushing
Pain as measured by PROMIS Pain Interference Short Form 8a | 12 weeks
  PROMIS Pain Interference Short Form 8a Questionnaire
Fatigue as measured by PROMIS Fatigue Short Form 8a | 12 weeks
  PROMIS Fatigue Short Form 8a Questionnaire
Grip Strength as measured by hand grip dynamometer | 12 weeks
  Participants exert as much force as possible using a Jamar hand grip dynamometer
Strength as measured by Biodex System 3 Multijoint dynamometer | 12 weeks
  Upper body strength is measured using a closed chain push/pull protocol. Lower body strength is measured using the knee flexion/extension protocol.
Balance as measured by the Timed Up and Go | 12 weeks
  The Timed to Up and Go test is performed using a chair with arms. The participants stand up from the chair, walk to a mark measured three meters from the chair then return back to the seat. A score of greater than or equal to 14 seconds (average) has been shown to indicate a high risk of falling.
Balance as measured by Biodex Limits of Stability | 12 weeks
  The Limits of Stability test is performed on the Biodex SD balance machine using the limits of stability protocol created by Biodex.
Balance as measured by Repeated Chair Stands | 12 weeks
  The repeated chair stands test is performed by asking participants to stand up and sit down 5 times as fast as possible. A score of greater than or equal to 14 seconds (average) has been shown to indicate a high risk of falling.
Walking velocity as measured by the GaitRite | 12 weeks
  20 meter walk is completed on the GaitRite mat

SECONDARY OUTCOMES:
Health Biomarkers as measured by blood analysis (insulin) | 12 weeks
  Participants undergo a fasted blood draw to assess insulin
Health Biomarkers as measured by blood analysis (lipids) | 12 weeks
  Participants undergo a fasted blood draw to assess lipids
Health Biomarkers as measured by blood analysis (fasting glucose) | 12 weeks
  Participants undergo a fasted blood draw to assess glucose
Anthropometric measurements (BMI) | 12 weeks
  height and weight are assessed to compute BMI
Circumference measurements to be reported as composite ratios (waist circumference, hip circumference, neck circumference) | 12 weeks
  circumference measures are completed at the neck, hip, and waist. Waist to hip ratios are computed (A/G ratio)
Physical Function with Mobility Aid as measured by PROMIS Physical Function with Mobility Aid 455b | 12 weeks
  PROMIS Physical Function with Mobility Aid 455b questionnaire
Anxiety as measured by PROMIS Emotional Distress-Anxiety Short Form 8a | 12 weeks
  PROMIS Emotional Distress-Anxiety Short Form 8a questionnaire
Depression as measured by PROMIS Emotional Distress-Depression Short Form 8a | 12 weeks
  PROMIS Emotional Distress-Depression Short Form 8a questionnaire
Sleep Disturbance as measured by PROMIS Sleep Disturbance Short Form 8a | 12 weeks
  PROMIS Sleep Disturbance Short Form 8a questionnaire
Ability to participate in social roles and activities as measured by PROMIS Ability to Participate in Social Roles and Activities Short Form 8a | 12 weeks
  PROMIS Ability to Participate in Social Roles and Activities Short Form 8a questionnaire
Nutrition Self-Efficacy as measured by the Nutrition Self-Efficacy Scale | 12 weeks
  Nutrition Self-Efficacy Scale
Physical Exercise Self-Efficacy as measured by the Physical Exercise Self Efficacy Scale | 12 weeks
  Physical Exercise Self Efficacy Scale
Pain intensity is measured by the PROMIS Pain Intensity Short Form | 12 weeks
  PROMIS Pain Intensity Short Form questionnaire
Body Composition as measured using a DEXA scan | 12 weeks
  GE Lunar Dual X-ray Absorptiometry is used to assess total body composition
Loneliness as measured by the Three-item loneliness scale | 12 weeks
  Three item loneliness scale

CONTACTS AND LOCATIONS:
Overall Officials: James Rimmer, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Lakeshore Foundation, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rimmer JH, Herman C, Wingo B, Fontaine K, Mehta T. Methodological and clinical implications of a three-in-one Russian doll design for tracking health trajectories and improving health and function through innovative exercise treatments in adults with disability. BMC Med Res Methodol. 2018 Mar 14;18(1):28. doi: 10.1186/s12874-018-0480-3. PMID 29540164